CLINICAL TRIAL: NCT00754260
Title: Caffeine Reduction Education And Overactive Bladder Symptoms
Brief Title: Caffeine Reduction and Overactive Bladder Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary Investigator left recruiting center.
Sponsor: University of New Mexico (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-277
Record Dates: First submitted 2008-09-02; First posted 2008-09-17 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caffiene reduction group (Experimental): Caffeine reduction group Intervention is to counseling to reduce caffeine intake
  Interventions: Behavioral: Caffeine reduction
- No caffeine reduction group (No Intervention): No Caffeine reduction group Intervention is to not counsel regarding caffeine intake

INTERVENTIONS:
Behavioral: Caffeine reduction — patients are randomized to receive caffeine reduction counseling versus no caffeine reduction counseling
  Arms: Caffiene reduction group

SUMMARY:
A. Statement of Objective: To conduct a randomized trial to evaluate the impact of caffeine restriction on Overactive Bladder(OAB) symptoms including urinary frequency, nocturia, incontinence episodes, symptom severity and bother and quality of life.

B. Specific Aims/Hypothesis:

1. To determine if reduction in caffeine intake decreases urinary frequency, nocturia and incontinence episodes as measured on a 3-day voiding diary in women with Overactive Bladder (OAB).

   We hypothesize that women with overactive bladder will report less frequent urination and decreased nocturia and incontinence episodes with caffeine reduction.
2. To determine whether caffeine reduction results in decreased symptom severity and bother and improved quality of life scores as measured by the Questionnaire for Incontinence Severity Index (ISI), Questionnaire for Urinary Incontinence Diagnosis (QUID), Urogenital Distress Inventory (UDI-6) and the Incontinence Impact Questionnaire (IIQ-7).

We hypothesize that women with OAB who reduce their intake of caffeine will report decreased symptom bother and improved quality of life as measured by the ISI, UDI-6 and the IIQ-

DETAILED DESCRIPTION:
Objective: To evaluate the impact of caffeine reduction education on urinary frequency.

Methods: Women with overactive bladder (OAB) symptoms who scored a 6 on the Questionnaire for Urinary Incontinence Diagnosis and who consumed at least 200 mg of caffeine daily were recruited. After completing baseline 3-day bladder diaries including amount and type of caffeine consumption, as well as validated urinary symptom severity, bother and quality of life questionnaires, women were randomized to receive caffeine reduction education vs. a control group who reviewed their voiding diary with no counseling to reduce caffeine; both groups were asked to maintain total fluid intake. Participants repeated the 3-day bladder diary and validated questionnaires following randomization. A total of 80 women were required to achieve 80% power with an alpha error of 0.05 to detect a difference of 1.3 in mean number of daily voids averaged over a 3-day voiding diary.

ELIGIBILITY:
Inclusion Criteria:

* only women 18 years and older with Overactive Bladder syndrome and who report that they consume an average of two cups of caffeinated beverages (approximately 200mg caffeine) daily will be included.

Exclusion Criteria:

* Women presenting with stress predominate bladder symptoms as evaluated by the QUID, urinary tract infection or hematuria as evaluated on urine dip analysis, currently pregnant or pregnant within the past six months or history of radiation to the pelvic floor will be excluded from participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2009-06-30 (Actual); Study Completion 2009-06-30 (Actual)

PRIMARY OUTCOMES:
urinary frequency, as measured on a 3-day voiding diary | baseline and 2 - 4 weeks

SECONDARY OUTCOMES:
Improved Quality of life scores | baseline and 2 - 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Rogers, Study Chair — University of New Mexico
Locations (2):
- United States (2):
  - Dr. Kammerer- Doak, Albuquerque, New Mexico
  - Tola Omotosho , MD, Albuquerque, New Mexico